CLINICAL TRIAL: NCT07154524
Title: Immunoadsorption for Treatment of Chronic Inflammatory Demyelinating Polyneuropathy (CIDP)
Acronym: IFTOC
Status: Recruiting | Type: Observational
Sponsor: University of Ulm (Other)
Collaborators: Fresenius Medical Care Deutschland GmbH (Industry)
Responsible Party: Principal Investigator, Albert Christian Ludolph, Prof., Prof. Dr., University of Ulm
Other Study IDs: IFTOC-2.21
Record Dates: First submitted 2025-08-27; First posted 2025-09-04 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-08

CONDITIONS: Chronic Inflammatory Demyelinating Polyneuropathy
Keywords: Chronic Inflammatory Demyelinating Polyneuropathy; Immunoadsorption; Long-term effects; therapy-refractory
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Immunoadsorption: Patients receiving Immunoadsorption as an escalation therapy after unsuccessful treatment with immunoglobulins or steroids

SUMMARY:
This study is designed as an explorative study aiming at exploring safety and efficacy of immunoadsorption (IA) in patients with Chronic Inflammatory Demyelinating Poly-neuropathy (CIDP) compared to intravenous immunoglobulins (IVIg) and methyl-prednisolone (MP). For this purpose, approximately 140 patients with CIDP will be included within the framework of the German multicenter network "Kompetenznetz Peripherer Nerv" (KKPNS).

The study will be purely observational. IA will be performed as an escalation therapy, i.e., in patients who did not respond to IVIg and/or MP treatment. Patients will be included in the study during ongoing IVIg or MP treatment and switched to IA during the 18-month observation period in case of an insufficient response. IA will be performed according to the therapeutic scheme of each participating center. A non-mandatory recommendation for number of sessions, treatment volumes, and frequency will be given (see below). Six-month follow-up visits including collection of standardized clini-cal data will be performed.

DETAILED DESCRIPTION:
Chronic inflammatory demyelinating polyneuropathy (CIDP) is a rare autoimmune-inflammatory disease which mainly affects the myelin sheaths of peripheral nerves, leading to paresis and sensory deficits.

Therapy of CIDP includes treatment with IVIg (evidence class Ia), MP (Ib), plasma exchange (PE; Ib), and various immunosuppressive drugs (IV). The European Federation of Neurological Societies (EFNS) guidelines recommend to begin with IVIg or MP as non-invasive options which are easy to apply, and to use PE in case of insufficient therapeutic response.

IA is a highly effective and well tolerated method to remove autoantibodies from the blood. Further proposed mechanisms of action include induction of autoantibody redistribution and subsequent immunomodulatory changes. During the procedure, the patient's plasma runs through adsorber systems which selectively bind human immunoglobulins before it is returned to the patient. Therefore, in contrast to PE, all other plasma proteins like coagulation factors are largely preserved, allowing higher treating frequencies and higher plasma volumes (PVs) to be processed. Adverse events in PE which are based on the loss of plasma proteins (like bleeding complications due to the loss of coagulation factors) are rare in IA, which is generally considered as a low-risk therapy. Furthermore, no substitution solutions like human albumin solutions or fresh frozen plasma are needed. Thus, better tolerability of IA compared to PE is regarded as one of the main advantages of IA and has been demonstrated in clinical studies. However, evidence for efficacy for IA in CIDP is low.

The objective of this trial is to investigate whether IA constitutes an effective and safe escalating therapeutic option in CIDP. For this purpose, IA will be performed in patients who showed insufficient therapeutic response to IVIg and/or MP, or who showed significant side effects under IVIG and/or MP therapy, and progression rates under therapy will be compared before and after the switch to IA.

One previous study in 20 patients8 found a higher response rate for patients treated with IA compared to PE (66.7% vs. 44.4%) after a follow-up of 4 weeks. Another non-randomized trial found that patients with therapy-refractory progressive disease courses could be stabilized by periodical cycles of IA9. However, in summary, evidence for the use of IA in CIDP is low, especially since there are no studies investigating the mid-term and long-term effects of repeated IA compared to other treatment options, and most studies refer to small sample sizes.

Therefore, in this study, we seek to evaluate safety and efficacy of IA in therapy-refractory CIDP in a prospective study design over a prolonged period of time, applying periodical cycles of therapies. Various standardized primary and secondary efficacy endpoints will be collected. The conduction within the German KKPNS network of specialized CIDP centers will facilitate the inclusion of 140 patients, enabling significantly higher evidence levels compared to pre-existing studies.

Objectives:

1. to investigate efficacy of IA measured by CIDP score and various other standardized efficacy parameters compared to a preceding IVIG and/or MP therapy.
2. to investigate safety of IA measured by type and frequency of Adverse Events (AEs) and Serious Adverse Events (SAEs) compared a preceding IVIG and/or MP therapy.
3. to investigate the effect of IA on various additional secondary endpoints, such as quality of life, compared to a preceding IVIg and/or MP therapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CIDP based on the EAN/PNS Guidelines on Diagnosis and Treatment of CIDP13
* age ≥ 18 years
* Willing and capable of giving written informed consent
* Currently receiving IVIg or MP treatment OR starting IVIg or MP treatment at baseline

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CIDP patients currently under treatment with immunoglobulins or steroids will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2025-08-27 (Actual); Primary Completion 2029-02-27 (Estimated); Study Completion 2029-08-27 (Estimated)

PRIMARY OUTCOMES:
Chronic Inflammatory Demyelinating Polyneuropathy (CIDP) Score | 18 months
  The CIDP score is a combined clinical score comprising the Inflammatory Neuropathy Cause and Treatment Score (INCAT), the Medical Research Council (MRC) and Vibrations Sensitivity Testing with a 256 Hz Ryder-Seiffel tuning fork. Range 0-480, higher values signify better outcome.

SECONDARY OUTCOMES:
Inflammatory Neuropathy Cause and Treatment Score (INCAT) | 18 months
  Range 0-10, higher values signify better outome
Medical Research Council (MRC) | 18 months
  Range 0-160; higher values signify better outcome. Musle power between 0/5 and 5/5 will be measured at 8 predifined muscle groups (agonist and antagonist, left and right, respectively) on upper and lower extrimities
Vibration Sensitivity | 18 months
  Vibration Sensitivity testing with a Ryder-Seiffel tuning fork
Inflammatory Rasch-built Overall Disability Scale (I-RODS) | 18 months
  Range 0-48; higher values signify better outcome
Overall Neuropathy Limitations Scale (ONLS) | 18 months
  Range 0-12, lower values signify better outcome
Pain Score (Visual Analog Scale) | 18 months
  Range 0-10, lower values signify better outcome
EuroQoL-5D-5L (EQ-5D-5L) | 18 months
Therapeutic Response | 18 months
  Share of patients with improvement of at least 1 point of INCAT
Type and frequency of Adverse Events (AEs) and Serious Adverse Events (SAEs) | 18 months
Neurofilament light chain (NfL) serum levels | 18 months
Paranodal antibody serum titers | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Dorst, Principal Investigator — University of Ulm
Locations (1):
- University of Ulm, Ulm, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Undecided